CLINICAL TRIAL: NCT03812432
Title: Near-infrared Fluorescence Cholecystocholangiography by Direct Intragallbladder Indocyanine Green Injection
Brief Title: Cholecystocholangiography by Direct Intragallbladder Injection of ICG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Son Espases (Other)
Responsible Party: Principal Investigator, F Xavier Molina Romero, MD PhD, Surgeon, Hospital Son Espases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMOL16012019
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- near-infrared cholecystocholangiography (Experimental): Each subject enrolled in this study will undergo near-infrared cholangiography fluorescence. Once the fundus is grasped and retracted, a needle-tipped cholangiogram catheter is introduced through the skin, adjacent to gallbladder. The catheter, guided by a grasping or dissecting instrument, is used to puncture the infundibulum of the gallbladder. Nine milliliters of bile is aspirated from the gallbladder into a syringe and and a indocianine green solution is injected into the gallbladder. The catheter is removed and the puncture site pinched closed with a grasper. Dissection is then performed under either ambient light or near-infrared mode. The surgical view of the gallbladder dissection is toggled back and forth between the two viewing.
  Interventions: Device: Near-infrared fluorescence cholecystocholangiography

INTERVENTIONS:
Device: Near-infrared fluorescence cholecystocholangiography — Device: Real-Time Fluorescence Imaging (VISERA ELITE II Imaging System). These device is used to identify anatomy, using infrared light that causes the indocianine green to fluoresce.

SUMMARY:
The objective of this clinical trial is to visualize the bile ducts by injecting a contrast that is only visible with infrared light. For this, a quantity of bile will be extracted from the gallbladder by puncture and the same amount of contrast will be introduced.

During the intervention teh tissue wil be exposure to infrared light to visualize the bile ducts. This technique aims to increase safety in surgery to avoid damaging bile or vascular structures during gallbladder interventions.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most commonly performed procedures in adult surgery. A rare but serious complication of laparoscopic cholecystectomy is bile duct injury, with a reported incidence of 0.3-1.5 %. Bile duct injury is often caused by misinterpretation of the anatomical structures rather than by insufficient technical skills. Generally, bile duct injury leads to bile leakage, causing abdominal sepsis. It can also lead to obstruction, with obstructive jaundice, eventually potentially leading to a need for liver transplantation in the worst case. Late recognition is common in bile duct injuries, resulting in significant morbidity and mortality, a lower quality of life and extra costs. A recent expert consensus report identified establishment of the critical view of safety as the single most important factor for overall safety during laparoscopic cholecystectomy. However, evidence suggests that surgeons may actually achieve this view far less often than they believe.

Numerous intraoperative visualization techniques and technologies have been developed to enhance the safety of laparoscopic cholecystectomy. There are mainly two intraoperative imaging techniques to consider: first, the historical X-ray-based intraoperative cholangiography, and secondly the emerging fluorescence-based intraoperative near-infrared cholangiography. Large retrospective and prospective studies have looked at the benefit of routine intraoperative radiographic cholangiography for detection of common bile duct stones and to identify or prevent bile duct injury. Whether this procedure should be performed routinely is still an active subject of debate as systematic reviews are inconclusive; however, several of the larger retrospective studies observed a decrease in frequency and severity of bile duct injury when intraoperative cholangiography is performed. Limiting factors for performing radiographic laparoscopic cholangiography include: it requires specific expertise in the technique and its interpretation; it involves the use of ionizing radiation; it is time-consuming; and it creates a risk for bile leakage and duct injury itself, since puncturing and cannulation of the cystic duct is required. These limitations justify the quest for alternative, less complicated techniques to visualize biliary anatomy during cholecystectomy. Fluorescence-based intraoperative near-infrared cholangiography during laparoscopic cholecystectomy has been introduced by Ishizawa et al. in recent years as a non-invasive, radiation-free, low-cost alternative for realtime visualization of the biliary anatomy. This technique requires near-infrared laparoscopic imaging systems, as well as the intravenous injection of a fluorophore, i.e., indocyanine green, which is eliminated through the biliary tree. Following exposure to the near-infrared fluorescenc light source, indocyanine green becomes fluorescent and highlights relevant biliary structures. Since the pioneer studies, a large number of trials have been conducted and several protocols are currently underway, in order to establish the clinical efficacy of near-infrared cholangiography. A recent systematic review of clinical studies on near-infrared cholangiography has reported high visualization rates of biliary structures, as a surrogate marker of clinical efficacy, before dissection of Calot's triangle. However, one of the most significant drawbacks of near-infrared cholangiography following systemic indocyanine green injection lies in the very high background signal due to the rapid accumulation of indocyanine green in the liver, which can impair the visualization of the biliary structures.

One of the strategies to improve the visualization of the cystic duct and the common bile duct, without suffering from the disturbing background liver enhancement, is to perform a near-infrared cholecystocholangiography, by injecting the fluorophore directly into the gallbladder, as previously demonstrated in a porcine experimental study.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for elective laparoscopic cholecystectomy.
2. Normal liver and renal function.
3. No hypersensitivity for iodine or indocianine green.
4. Able to understand nature of the study procedures.
5. Willing to participate and with written informed consent.

Exclusion Criteria:

1. Age < 18 years.
2. Liver or renal insufficiency.
3. Known iodine or indocianine green hypersensitivity.
4. Pregnancy or breastfeeding.
5. Not able to understand nature of the study procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visualization of the cystic duct, common hepatic duct, common bile duct and cysticocholedochal junction. | Intra-operatively
  Percentage of patients for whom fluorescence allows visualize cystic duct, common hepatic duct, common bile duct and cysticocholedochal junction with precision. cysticocholedochal junction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands, Spain